CLINICAL TRIAL: NCT07206849
Title: A Phase 2 Study of Tovorafenib in Pediatric and Young Adult Patients Newly Diagnosed With High-Grade Glioma (HGG), Including Diffuse Intrinsic Pontine Glioma (DIPG), Which Harbor Alterations in the Mitogen-Activated Protein Kinase (MAPK) Pathway
Brief Title: Study of Tovorafenib in High-Grade Glioma and Diffuse Intrinsic Pontine Glioma (DIPG)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONNECT TarGeT-B; R01FD008167 (FDA)
Record Dates: First submitted 2025-09-18; First posted 2025-10-03 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-09

CONDITIONS: High Grade Glioma (HGG) of the Brain With BRAF Aberration; High Grade Glioma (III or IV); Diffuse Intrinsic Pontine Glioma; High Grade Glioma; WHO Grade 3 Glioma; WHO Grade 4 Glioma; Metastatic Brain Tumor
Keywords: tovorafenib; high grade glioma
MeSH Terms: conditions — Glioma; Diffuse Intrinsic Pontine Glioma; Brain Neoplasms | interventions — tovorafenib

STUDY DESIGN:
Intervention Model Description: Tovorafenib
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Stratum A - localized HGG (Experimental): Patients with intracranial, localized, non-pontine, and non-thalamic HGG harboring a BRAFV600 mutation (who do not meet criteria for Strata B or C).
  Interventions: Drug: Tovorafenib
- Stratum B - DIPG (Experimental): Patients with DIPG/DMG as defined in Section 4.1.3 OR patients with localized, non-pontine, non-thalamic HGG harboring a MAPK alteration not included in Stratum A (KIAA1549:BRAF fusion, KRAS/NRAS, CRAF/RAF1, other RAF mutation, or FGFR alteration) OR patients with primary spinal tumors.
  Interventions: Drug: Tovorafenib
- Stratum C - metastatic HGG (Experimental): Patients with metastatic HGG (including metastatic DIPG/DMG) harboring a MAPK alteration (BRAFV600, KIAA1549:BRAF fusion, KRAS/NRAS, CRAF/RAF1, other RAF mutation, or FGFR alteration).
  Interventions: Drug: Tovorafenib

INTERVENTIONS:
Drug: Tovorafenib — Tovorafenib will be given orally once weekly (QW) throughout each cycle.

SUMMARY:
The goal of this study is to determine the efficacy of the study drugs tovorafenib to treat pediatric and young adult patients newly diagnosed with a high-grade glioma (HGG), including DIPG, that have genetic changes in pathways (MAPK) that this drug targets.

The main question the study aims to answer is whether tovorafenib can prolong the life of patients diagnosed with HGG, including DIPG.

DETAILED DESCRIPTION:
In this phase 2 study, pediatric, adolescent, and young adult patients with newly-diagnosed HGG and DIPG harboring alterations in the MAPK pathway will be treated with tovorafenib following initial standard-of-care treatment with radiotherapy (RT). The objectives of the trial are to assess the progression free survival (PFS) and overall survival (OS) distribution for patients with newly diagnosed HGG. This trial will include three strata. Stratum A will evaluate PFS and OS in newly diagnosed patients with HGG harboring a BRAFV600 mutation. Stratum B will evaluate PFS and OS in newly- diagnosed patients with DIPG/DMG, primary spinal cord HGG with MAPK alterations, and other MAPK alterations will be descriptively analyzed. In Stratum C, metastatic patients will be assessed for feasibility of treatment with tovorafenib post craniospinal irradiation. Tovorafenib has previously been studied in pediatrics. The recommended pediatric dosing of tovorafenib is 380mg/m2 every week (QW) and will be used as the starting dose in all strata of this study. We hypothesize that tovorafenib will improve PFS in newly-diagnosed HGG.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have previously enrolled on TarGeT-SCR.

  1. Age Patients must be ≥12 months and ≤39 years of age at the time of enrollment on TarGeT-SCR.
  2. Body Surface Area (BSA) Patients must have a BSA >0.3m2.
  3. Diagnosis:

     * Patients with a newly-diagnosed HGG, including DIPG, which harbor alterations in the MAPK pathway are eligible. All patients must have tumor tissue from diagnostic biopsy or resection. The diagnosis of HGG, including DIPG, must have been confirmed through TarGeT-SCR.
     * For the diagnosis of DIPG, patients must have a tumor with pontine epicenter and diffuse involvement of at least 2/3 of the pons, with histopathology consistent with diffuse WHO Grade 2-4 glioma.
     * All other HGGs must be WHO Grade 3 or 4.
  4. Disease Status

     • Patients must be newly diagnosed and enroll and start treatment within 35 days of completion of radiotherapy.

     • Measurable disease is not required. Patients without measurable disease are eligible.
     * Patients with primary spinal tumors are eligible.
     * Patients with secondary or radiation-induced HGG are eligible.
  5. TarGeT-B Strata Definitions

     Patients must be able to be assigned to one of the strata below:

     • Stratum A: Patients with intracranial, localized, non-pontine, and non-thalamic HGG harboring a BRAFV600 mutation (who do not meet criteria for Strata B or C).
     * Stratum B: Patients with DIPG/DMG as defined in Section 4.1.3 OR patients with localized, non-pontine, non-thalamic HGG harboring a MAPK alteration not included in Stratum A (KIAA1549:BRAF fusion, KRAS/NRAS, CRAF/RAF1, other RAF mutation, or FGFR alteration) OR patients with primary spinal tumors.
     * Stratum C: Patients with metastatic HGG (including metastatic DIPG/DMG) harboring a MAPK alteration (BRAFV600, KIAA1549:BRAF fusion, KRAS/NRAS, CRAF/RAF1, other RAF mutation, or FGFR alteration).
  6. Presence of at least one relevant actionable somatic alteration:

     • MAPK pathway alteration(s): BRAFV600 mutation (Strata A or C)
     * KIAA1549:BRAF fusion (Strata B or C)
     * KRAS/NRAS alteration (Strata B or C)
     * CRAF/RAF1 alteration (Strata B or C)
     * other RAF mutations (Strata B or C)
     * FGFR alteration (Strata B or C)
  7. Performance Level:

     Karnofsky ≥ 50 for patients > 16 years of age and Lansky ≥ 50 for patients ≤ 16 years of age (Appendix I). Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
  8. Prior Therapy for HGG:

     o Surgery, radiation (RT), and/or dexamethasone are permissible. Temozolomide administered concurrently with RT is permissible but discouraged for patients with DIPG/DMG. No other prior anticancer therapy for HGG will be allowed.

     o Radiation therapy requirements: Patients must have received photon or proton focal radiotherapy if enrolling on Stratum A or B. Patients must have received craniospinal irradiation if enrolling on Stratum C.

     o Radiotherapy, delivered photon or proton beam, must have been administered at a standard dose, including:

     o 54 Gy in 30 fractions for DIPG

     o 54-59.4 Gy in 30-33 fractions for other HGG

     o 45-54 Gy for primary spinal cord HGG

     o And/or 36-39.6 Gy craniospinal for patients with spinal or leptomeningeal metastatic disease with supplemental boost to 45-54 Gy for metastasis within the thecal sac and 54-60 Gy for intracranial metastasis.

     o Any variances in the radiotherapy dose within 10% of standard doses outlined above will be discussed with the Sponsor-Investigator to confirm eligibility prior to study enrollment.

     o Timing between diagnosis and start of RT: Patients must have started RT within 31 calendar days of initial diagnosis which is defined as the date of diagnostic biopsy or resection. If a patient underwent two upfront surgeries e.g., biopsy then resection or debulking, this is the date of the second surgery.
     * Timing post-RT: Patients must enroll and start treatment on TarGeT-B no later than 35 calendar days post-completion of RT. The earliest patients can begin protocol treatment is 28 calendar days post-completion of RT.
  9. Organ Function Requirements
* Adequate Bone Marrow Function Defined as:

  • Peripheral absolute neutrophil count (ANC) >= 1000/mm3.

  • Platelet count >= 100,000/mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment).

  • Hemoglobin >8 g/dL (may be transfused).
* Adequate Renal Function Defined as:

Creatinine clearance or radioisotope GFR > 70ml/min/1.73 m2 OR serum creatinine based on age/gender as follows:

Maximum Serum Creatinine (mg/dL) Age Male Female 1 to < 2 years 0.6 0.6 2 to < 6 years 0.8 0.8 6 to < 10 years 1 1 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.4

* 16 years 1.7 1.4 The threshold creatinine values in this table were derived from the Schwartz formula for estimating GFR (Schwartz et al. J. Peds, 106:522, 1985) utilizing child length and stature data published by the CDC.

  * Adequate Liver Function Defined as:

    * Total bilirubin ≤ 1.5 times institutional upper limit of normal (ULN).
    * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 3 times the ULN.
    * Serum albumin ≥ 2g/dL.
  * Adequate Cardiac Function Defined as:

    • Left Ventricular Ejection fraction of ≥ 50% as measured by echocardiogram or multiple-gated acquisition (MUGA).
    * QTc ≤ 450 msec (by Bazett formula).
  * Adequate Neurologic Function Defined as:

    * Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled (see Appendix II).
  * Normal Thyroid Function Defined as:

    • Free throxine (T4) within institutional guidelines for normal range. It is acceptable for patient to be on thyroid supplementation as long as free T4 is within institutional guidelines for normal range prior to starting treatment.

    10) Informed Consent All patients and/or their parents or legally authorized representatives must sign a written Informed Consent and Assent, when appropriate, will be obtained according to institutional guidelines.

Exclusion Criteria:

1. Pregnancy or breastfeeding.
2. Other Exclusion Criteria

   • Patients with neurofibromatosis type 1 (NF-1) are not eligible for this study.

   • Infection: Patients who have an uncontrolled infection are not eligible.

   • Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study are not eligible.

   • Patients with uncontrolled GI disease or other condition that could affect absorption or predispose participant to gastrointestinal ulceration are not eligible.
3. Concomitant Medications • Corticosteroids: Patients receiving corticosteroids are eligible, but the use of corticosteroids must be reported.

   • Investigational Agents/Drugs: Patients who are currently receiving another investigational drug are not eligible. This includes targeted agents, monoclonal antibodies, herbal supplements, or other investigational agents other than tovorafenib.

   • Anti-cancer Agents: Patients who are currently receiving other anti-cancer agents are not eligible with the exception of temozolomide given concurrently with radiotherapy.

   • Anticonvulsants: Patients who are receiving enzyme-inducing anticonvulsants as listed in Appendix II, are not eligible.

   • Patients who are receiving medications known to prolong QTc interval as listed in Appendix III are not eligible.

   • As tovorafenib is a substrate of CYP2C8, patients should not take strong inhibitors or inducers of CYP2C8 (See Appendix VI), as they could alter the drug's pharmacokinetics. Medications that are substrates of CYP2C8 or CYP3A4 are allowed but should be used with caution.

   • Medications that are substrates of breast cancer resistance protein (BCRP) with a narrow therapeutic index are prohibited during this study (Appendix IV).
   * Patients who are receiving duloxetine, alosetron, or theophylline (CYP1A2 inhibitors) are not eligible.
   * Patients on beta-blockers are not eligible.
   * Selective serotonin reuptake inhibitors (SSRIs) such as citalopram (Celexa), escitalopram (Lexapro), Fluoxetine (Prozac), fluvoxamine (Luvox), paroxetine (Paxil), sertraline (Zoloft) should be used with caution but are not contraindicated.
   * Anticoagulants: patients who are receiving therapeutic anticoagulants including warfarin, low-molecular weight heparin are not eligible.

5) Patients with prior or ongoing clinically significant medical or psychiatric condition that, in the investigator's opinion, could affect the safety of the participant, or could impair the assessment of study results are not eligible.

Ages: 12 Months to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 79 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2030-03-01 (Estimated); Study Completion 2037-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival Stratum A | 6 years
  Estimate the progression-free survival (PFS) distribution for pediatric and young adult patients (age: ≥12 months and ≤39 years) with newly-diagnosed BRAFV600 mutant HGG (Stratum A) who receive tovorafenib monotherapy post RT compared to molecularly-stratified, matched historical controls.

SECONDARY OUTCOMES:
Overall Survival Stratum A | 6 years
  Estimate the overall survival (OS) distribution for pediatric and young adult patients with newly-diagnosed BRAFV600 mutant HGG (Stratum A) who receive tovorafenib post RT compared to molecularly-stratified, matched historical controls.
OS Stratum B | 6 years
  Describe OS for pediatric and young adult patients newly diagnosed with DIPG or DMG harboring MAPK pathway alterations who receive tovorafenib post RT (Stratum B).
PFS Stratum B | 6 years
  Describe PFS for pediatric and young adult patients newly diagnosed with HGG harboring MAPK alterations not included in Stratum A who receive tovorafenib post RT (Stratum B).
OS Stratum B | 6 years
  Describe the OS for pediatric and young adult patients newly diagnosed with primary spinal cord HGG harboring a MAPK alteration who receive tovorafenib post RT (Stratum B).
Establish the RP2D of tovorafenib - Stratum C | At the end of Cycle 1 (each cycle is 28 days)
  Evaluate the feasibility of administration of tovorafenib post craniospinal RT in pediatric and young adult patients with newly diagnosed, metastatic HGG harboring a MAPK alteration (Stratum C).
OS Stratum C | 6 years
  Describe OS for pediatric and young adult patients with newly-diagnosed, metastatic HGG who receive tovorafenib post RT (Stratum C).
ORR | 6 years
  Evaluate the radiographic objective response rate (ORR [complete response (CR) + partial response (PR)]) to tovorafenib treatment post RT in pediatric and young adult patients with newly diagnosed HGG and DIPG/DMG that harbor MAPK alterations (all Strata).
Number of participants with tovorafenib-related adverse events as assessed by CTCAE v5.0 | From Day 1 of protocol treatment through 30 days following end of protocol treatment
  Assess and further characterize the safety and toxicity of post-RT tovorafenib in pediatric and young adult patients newly diagnosed with HGG, including DIPG. This will be achieved by calculating the number of participants with, as well as frequency and severity of, tovorafenib-related Adverse Events as assessed by CTCAE v5.0.
Correlation between genomic status, recurrence, radiographic response | 6 years
  Explore longitudinal associations of genomic, transcriptomic, epigenetic, and/or immunologic alterations of tumor at diagnosis, recurrence, or autopsy with radiographic response, advanced neuro-imaging measures, and patient-reported outcomes.
Evaluate Health-Related Quality of Life Outcomes | 6 years
  Evaluate health-related quality of life outcomes of pediatric and young adult patients newly-diagnosed with HGG, including DIPG, treated with tovorafenib, by patient and/or parent reporting at key timepoints in therapy using the patient reported outcomes measurement information system (PROMIS) survey which will be completed by consenting participants every other cycle for the length of their treatment (all Strata).
PFS Stratum B | 6 years
  Describe the PFS for pediatric and young adult patients newly diagnosed with primary spinal cord HGG harboring a MAPK alteration who receive tovorafenib post RT (Stratum B).
PFS Stratum C | 6 years
  Describe PFS for pediatric and young adult patients with newly-diagnosed, metastatic HGG who receive tovorafenib post RT (Stratum C).

IPD SHARING:
Plan to Share IPD: No